CLINICAL TRIAL: NCT06193629
Title: A Multicenter, Double-blind, Placebo-randomized Controlled Clinical Study on the Treatment of Non-alcoholic Steatohepatitis With Tibetan Drug Langqing Atar
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shupei Li (Other)
Responsible Party: Sponsor-Investigator, Shupei Li, student, Jinling Hospital, China
Organization: Jinling Hospital, China (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: DZQH-KYLLFS-23-25
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: NASH

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lang Qingata (Experimental): Lang Qingata: (Artificial bezoar: 0.1g, Safflower: 15g, five spirit fat: 15g, Tangerine: 30g, Swertia: 15g, nutmeg: 10g, Astragalus: 25g, wood fragrance: 10g, Parasol tiger grass: 15g, Coriander fruit: 10g, Agarwood: 3g, pomegranate seed: 20g, Rhododendron: 8g, Dongquai fruit: 15g, licorice: 10g). Water decoction (hospital decoction), Decoction in water for oral use，2 times/day, 4 weeks for a course of treatment.
  Interventions: Drug: Lang Qingata
- placebo group (Placebo Comparator): Placebo is a Chinese medicine granule with 5% active ingredient and has the same taste as Lang Qingata，Decoction in water for oral use。
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Lang Qingata — Lang Qingata: (Artificial bezoar: 0.1g, Safflower: 15g, five spirit fat: 15g, Tangerine: 30g, Swertia: 15g, nutmeg: 10g, Astragalus: 25g, wood fragrance: 10g, Parasol tiger grass: 15g, Coriander fruit: 10g, Agarwood: 3g, pomegranate seed: 20g, Rhododendron: 8g, Dongquai fruit: 15g, licorice: 10g). Water decoction (hospital decoction), Decoction in water for oral use，2 times/day, 4 weeks for a course of treatment.
  Arms: Lang Qingata
Drug: placebo — Placebo is a Chinese medicine granule with 5% active ingredient and has the same taste as Lang Qingata，Decoction in water for oral use
  Arms: placebo group

SUMMARY:
non-alcoholic steatohepatitis (NASH) is an inflammatory liver disease caused by the accumulation of fat in liver cells. With the change of living habits and diet, the incidence of Nash continues to increase. In the early stage, NASH generally has no obvious symptoms. With the progression of the disease and the aggravation of liver damage, it may induce fatigue, loss of body mass, and pain in the right upper abdomen, which seriously affects the health of patients. There are no specific drugs to treat NASH in clinical practice. Increasing exercise, taking drugs to avoid liver damage, controlling diet and other methods can alleviate clinical symptoms to a certain extent, but the stability of disease control is poor, and it is easy to develop into cirrhosis, threatening the life safety of patients. However, there are few clinical reports on the effect of drugs on NASH. In the previous treatment of patients with liver fibrosis, our research group found that non-alcoholic steatohepatitis NASH induced liver fibrosis has a good effect, suggesting that Langqingata may improve NASH. Based on this, this study observed the total effective rate of Lang Qingata in the treatment of nonalcoholic steatohepatic NASH.

DETAILED DESCRIPTION:
Scheme introduction

1. Test purpose A multi-center, prospective, double-blind, placebo-randomized controlled clinical trial was conducted to observe the total effective rate of Lang Qingata (observation group) and placebo (control group) through drug intervention in patients with nonalcoholic steatohepatitis, providing evidence for the treatment of patients with nonalcoholic steatohepatitis.
2. Research the overall design 2.1 Overall design of the experiment Multicenter, prospective, double-blind, placebo-randomized controlled clinical trial.

   2.2 Enrolled cases Patients ≥18 years of age and ≤60 years of age who meet the diagnostic criteria for NASH.

   2.3 Basis for calculation of test sample size The study was a randomized, double-blind, placebo-controlled multicenter clinical study with overall clinical efficacy as the primary endpoint. According to previous research reports, the estimated effective rate of the placebo group was 50%, and the previous study of our group suggested that the effective rate of Lang Qingata was no less than 70%. Chi-square test will be used to compare the effective rate of the two groups (H0: π experimental group =π control group, H1: π experimental group ≠π control group), the test level α=0.05 (bilateral), the certainty is 80%, the sample size ratio of the experimental group and the control group is 1:1, assuming that the shedding rate is not more than 10%. According to the above parameters, the total sample size was estimated by PASS software to be 150 cases, including 75 cases in the experimental group and 75 cases in the control group.

   2.4 Case grouping and case distribution plan Eligible subjects were assigned to Lang Qingata group and placebo group in a ratio of 1:1. Each group was intended to include 75 patients.

   2.5 Random allocation Method A block randomization scheme was adopted, which was implemented based on the eRand Central Randomization system of clinical trials, and all centers competed for inclusion.
3. Diagnostic criteria 3.1 Diagnostic criteria for NASH in Western medicine:

(1) No history of alcohol abuse, that is, alcohol content < 30 g/d for men and < 20 g/d for women.

(2) Exclude some diseases associated with NASH, such as drug-induced liver disease, autoimmune liver disease, and total parenteral nutrition. (3) Clinical symptoms include fatigue, poor digestion, liver pain, liver and spleen enlargement, and there may be no significant symptoms.

(4) In patients with recent body mass gain and/or metabolic syndrome-related manifestations, unexplained serum ALT and/or AST and GGT continued to increase for more than six months; (5) Liver color ultrasound or CT meets the diagnostic criteria for diffuse fatty liver disease, and no other cause can be explained.

3.2 TCM diagnostic criteria of this study Refer to the Consensus Opinion on the Diagnosis and Treatment of Integrative Chinese and Western Medicine for Non-alcoholic Fatty Liver Disease (2017).

Syndrome of liver depression and spleen deficiency:

Main symptoms :(1) hypochondrium distension; (2) bitter and dry mouth; (3) Formed stool or loose stool; (4) fatigue and fatigue; Secondary symptoms :(1) loss of appetite; (2) Abdominal distension discomfort; (3) upset insomnia; (4) sweating; (5) Unfavorable urination; Tongue and pulse: light red tongue, thin white or white tongue coating, teeth marks, fine pulse string.

Syndrome type determination: with 2 or more main symptoms and 1 or more secondary symptoms, refer to tongue and pulse.

3.3. CT diagnostic criteria The density of normal liver was higher than that of spleen, that is, liver/spleen CT value was > 1. Mild fatty liver :0.7 < liver/spleen CT value ≤1.0; Moderate fatty liver :0.5 < liver/spleen CT value ≤0.7; Severe fatty liver: liver/spleen CT value < 0.5.

3.4 BMI diagnostic criteria The normal range of body mass index (BMI) was 18.5-23.9kg/m². Between 24.0 and 27.9kg/m² indicates overweight, and ≥28.0kg/m² indicates obesity.

3.5 Liver color ultrasound diagnostic criteria Those who meet items (1) and (2)-(4) below are diagnosed as mild fatty liver; Those who meet the two items (1) and (2)-(4) below are diagnosed with moderate fatty liver; Those who meet items (1), (2)-(4) and (5) below are diagnosed with severe fatty liver disease.

1. The front field echo of liver was enhanced, the echo was stronger than that of kidney and spleen, and the far field echo was attenuated;
2. The intrahepatic duct structure is blurred;
3. The liver is enlarged and full, and the edges and corners are blunted;
4. The intrahepatic color blood flow signal is reduced or not easy to show, but the intrahepatic blood vessels are normal;
5. The echo display of the right lobe capsule and transverse septum of the liver was unclear or incomplete.

4. Case selection 4.1 Inclusion criteria

1. Signed written informed consent;
2. Age 18-60 years old, gender is not limited;
3. Meet the clinical diagnostic criteria for NASH (see study Content 3 diagnostic criteria);
4. The subjects could follow the follow-up plan, objectively describe the symptoms, and cooperate with the completion of the scale;
5. Non-lactating pregnant women and no pregnancy plan during the test;
6. Do not participate in any clinical trials for 3 months before and during the trial.

4.2 Exclusion Criteria

1. < 18 years old or > 60 years old;
2. People who are allergic or allergic to the ingredients of this medicine;
3. Liver cirrhosis and liver tumor patients or ALT, AST≥ 5 times the normal upper limit, liver function damage is more serious This;
4. Women who are pregnant, breastfeeding or planning to become pregnant during the trial;
5. Complicated with viral hepatitis, alcoholic hepatitis, autoimmune liver disease and cirrhosis, liver cells Patients with other liver diseases such as cancer, serious heart, brain, and kidney diseases, such as chronic cardiac insufficiency;
6. suffering from other serious diseases, such as tumors and other special blood diseases;
7. Poor compliance, unable to cooperate with the completion of the experiment. 4.3 Exclusion Criteria

1) After inclusion, it is found that they do not meet the inclusion criteria or meet any exclusion criteria and are mistakenly included; 2) Can not tolerate or fail to carry out drug intervention on time; 3) Subject withdraws informed consent. 4.4 Exit Standards and Procedures 4.4.1 Exit Standard

1. The subjects voluntarily withdrew from the trial: they felt that the efficacy was not good, they felt that some adverse events were difficult to tolerate, and they lost follow-up for unknown reasons.
2. The investigator decides to withdraw from the trial:

   1. If the risk/benefit ratio is found to be unacceptable for the subject, the investigator or secondary investigator has the right and responsibility to discontinue treatment of the subject.
   2. If factors beyond the investigator's control significantly affect the course of the trial and/or the interpretation of the trial results, the investigator must discontinue treatment of the subject.
3. If any of the following occurs, the subject must withdraw from the test:

   1. Subject or his legal representative withdraws informed consent.
   2. Adverse events that occur should be withdrawn from the clinical trial as determined by the physician.

4.4.2 Exit Procedure Subjects may withdraw from the trial at any time and for any reason. The researchers discontinue the subjects' treatment, and the discontinuation is "permanent"; once a subject drops out, he or she will not be allowed back into the study. From the moment the subject withdraws the informed consent, the subject may no longer be contacted directly to obtain new information (including the data query clarification form).

Collect at least the following information when the subject withdraws:

1. Reasons for exit;
2. The date and time of the last assessment and/or contact. Arrange an appropriate visit (telephone or outpatient review);
3. (serious) adverse events;
4. Final evaluation. Every effort must be made to ensure that all test processes and evaluations of the last visit plan are carried out.

If a subject withdraws before a drug intervention, the subject will not be included in the efficacy and safety analysis. If the subject withdraws after the medication intervention, all available data will be accounted for in the efficacy and safety analysis.

4.5 Criteria for discontinuation of tests

1. Serious adverse events related to the drug intervention occurred during the trial.
2. Significant errors in the clinical trial protocol were found in the trial, making it difficult to evaluate the drug intervention.
3. If the designed scheme in the experiment has major deviations in the implementation, it is difficult to evaluate the main observation indicators if it is continued.
4. The sponsor requests suspension (such as funding reasons, management reasons, etc.).

5. Clinical trial procedure 5.1 Overview We will screen qualified patients according to uniform norms for inclusion, and improve the initial assessment examination and informed consent signature before patients are enrolled. Patients were assigned to Langqingata or placebo using an envelope randomization assignment tool. After random allocation, the subjects received drug intervention within the prescribed time, and the subjects were asked to receive regular telephone follow-up or outpatient follow-up, receive imaging examination, laboratory examination and other assessment of the condition, and collect complete medical history data for statistics.

5.2 Screening of qualified patients In principle, the subject's written informed consent must be obtained before any trial related procedure can be performed. After informed consent is obtained, the researchers responsible for data collection obtain the grouping information through the envelope.

5.3 Preoperative, intraoperative and postoperative treatment

1. Preparation before treatment:

   Patients in the treatment group and the control group, on the basis of normal medication, corrected their bad lifestyle, optimized their diet structure, limited the intake of high-sugar and high-fat diets, increased the proportion of high-fiber diets such as vegetables, beans and fruits, avoided drinking alcohol as much as possible, exercised moderately, strengthened weight control, avoided overwork, and paid attention to rest.

   Before drug intervention, subjects were assessed for weight and height, and blood samples were obtained for routine biochemical tests of liver function (ALT, AST, GGT), lipid levels (TG, TC, HDL-C, LDL-C), fasting glucose FPG, and inflammatory factors (TNF-α, IL-1β, IL-6). The activities of MDA and SOD were analyzed qualitatively by B-ultrasound and quantitatively by CT values of liver/spleen.
2. Treatment group:

The enrolled patients were randomly divided into two groups:

1. Lang Qingata: (artificial bezoar: 0.1g, Safflower: 15g, five Lingzhi: 15g, Tangerine: 30g, Swertia: 15g, nutmeg: 10g, Astragalus: 25g, wood fragrance: 10g, Parasol tiger grass: 15g, coriander fruit: 10g, Agarwood: 3g, pomegranate seed: 20g, Rhododendron: 8g, Dongquai fruit: 15g, licorice: 10g). Water decoction (hospital decoction), 2 times/day, 4 weeks for a course of treatment.
2. Placebo group :2 times/day, 4 weeks for one course. 3) Post-treatment: Both groups were treated for 2 months. Subjects were followed up at 2, 4 and 8 weeks, respectively, and the therapeutic effect was evaluated after the treatment was completed.

6. Observation indicators and judgment criteria 8 weeks was used as the end point of follow-up, and the last follow-up was used as the end point of follow-up for those who dropped out of the trial.

Total effective rate of clinical effect = (cure + obvious + effective) cases/total cases ×100%.

6.1 Observation Indicators 6.1.1 Main observation indicators To observe the total effective rate of Lang Qingata in the treatment of nonalcoholic steatohepatic NASH 6.1.2 Minor Observation Indicators A: Body mass index (BMI) before and after treatment B: Ultrasound before and after treatment C: Liver function before and after treatment (ALT, AST, GGT, ALP) D: Blood lipid levels before and after treatment (TG, TC, HDL-C, LDL-C, TBIL) E: Inflammatory cytokines (TNF-α, IL-1β, IL-6) before and after treatment F: CT values of liver/spleen before and after treatment G: Fasting blood glucose FPG before and after treatment H: MDA and SOD activity before and after treatment I: TCM syndrome scores before and after treatment are scored by two associate chief physicians (see Attached Table 1 and Attached Table 2) 6.2Comprehensive efficacy criteria: According to the 2002 "Guiding Principles for Clinical Research of New Chinese Medicine" and literature.

Cure: Clinical symptoms completely disappeared, liver echo by B-ultrasound basically returned to normal, liver/spleen CT fatty liver features disappeared, liver enzymology (ALT, AST, GGT) and blood lipid (TC, TG, HDL-C, LDL-C) indicators returned to normal; Obvious effect: The clinical symptoms disappeared basically or completely, the liver echo disease grade of B-ultrasound examination decreased by 2 grades, the fatty liver disease grade of liver/spleen CT decreased by 2 grades, ALT and (or)AST and GGT decreased by >50%, and the improvement of blood lipids met any of the following criteria :TC decreased by ≥20%, TG decreased by ≥40%. HDL-C increased ≥0.26mmol/L; Effective: Clinical symptoms improved significantly, liver echo disease grade in B-ultrasound examination decreased by 1 grade, fatty liver disease grade in liver/spleen CT decreased by 1 grade, 30% < ALT and (or)AST and GGT decreased by < 50%, blood lipid improvement met any of the following criteria :TC decreased by ≥10% but < 20%, TG decreased by ≥20% but < 40%. HDL-C increased ≥0.13mmol/L but < 0.26mmol/L Ineffective: Clinical symptoms and test results do not meet the above criteria.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria: Participants must meet all of the following criteria to enter the trial.

  1. Signed written informed consent;
  2. Age 18-60 years old, gender is not limited;
  3. Meet the clinical diagnostic criteria for NASH; (See study content 3 Diagnostic criteria)
  4. The subjects could follow the follow-up plan, objectively describe the symptoms, and cooperate with the completion of the scale;
  5. Non-lactating pregnant women and no pregnancy plan during the test;
  6. Do not participate in any clinical trials for 3 months before and during the trial.

Exclusion Criteria:

1. < 18 years old or > 60 years old;
2. People who are allergic or allergic to the ingredients of this medicine;
3. Liver cirrhosis and liver tumor patients or ALT, AST≥ 5 times the normal upper limit, liver function damage is more serious This;
4. Women who are pregnant, breastfeeding or planning to become pregnant during the trial;
5. Complicated with viral hepatitis, alcoholic hepatitis, autoimmune liver disease and cirrhosis, liver cells Patients with other liver diseases such as cancer, serious heart, brain, and kidney diseases, such as chronic cardiac insufficiency;
6. suffering from other serious diseases, such as tumors and other special blood diseases;
7. Poor compliance, unable to cooperate with the completion of the experiment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The total effective rate of Lang Qing Atta in the treatment of nonalcoholic steatohepatic NASH | 2month
  Total effective rate of clinical effect = (cure + obvious + effective) cases/total cases
  ×100%.The criteria for cure, efficacy, and effectiveness are described in the study

SECONDARY OUTCOMES:
BMI | 2month
  Body mass index (BMI) before and after treatment
B-ultrasound | 2month
  B-ultrasound before and after treatment
AST change from baseline | 2month
  Changes in aspartate aminotransferase (AST) relative to baseline in the treatment group at week 8 visit were summarized
Blood lipid levels | 2month
  Blood lipid levels (TG, TC, HDL-C, LDL-C, TBIL) before and after treatment
Inflammatory cytokines | 2month
  Inflammatory cytokines (TNF-α, IL-1β, IL-6) before and after treatment
CT values of liver/spleen | 2month
  CT values of liver/spleen before and after treatment
Fasting blood glucose FPG | 2month
  Fasting blood glucose FPG before and after treatment
TCM syndrome integral | 2month
  The TCM syndrome score before and after treatment is scored by two associate chief physicians
ALT change from baseline | 2month
  Changes in aspartate aminotransferase (ALT) relative to baseline in the treatment group at week 8 visit were summarized
GGT change from baseline | 2month
  Changes in aspartate aminotransferase (GGT) relative to baseline in the treatment group at week 8 visit were summarized
ALP change from baseline | 2month
  Changes in aspartate aminotransferase (ALP) relative to baseline in the treatment group at week 8 visit were summarized

CONTACTS AND LOCATIONS:
Locations (1):
- A multicenter, double-blind, placebo-randomized controlled clinical study on the treatment of non-alcoholic steatohepatitis with Tibetan drug Langqing Atta, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No